CLINICAL TRIAL: NCT05410574
Title: Family-Based Behavioral Treatment for Childhood Survivors of Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient staff
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202205124
Record Dates: First submitted 2022-05-24; First posted 2022-06-08 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Overweight/obesity; Weight management; Family based behavioral weight loss treatment (FBT)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children: Family-based Behavioral Weight Loss Treatment (FBT) (Experimental): * Traffic Light Eating Plan: All foods are assigned a color of the traffic light depending on their energy density & nutritional quality. Participants are encouraged to set dietary goals to decrease the number of RED food servings consumed daily & to increase the consumption of GREEN & YELLOW foods.
  * Traffic Light Activity Plan: Activities are assigned colors of the traffic light depending on intensity levels. Families are encouraged to increase time spent in GREEN activities and decreased RED activities.
  * Behavior Change Strategies: Behavior modification will be fostered using several different strategies
  * Social Facilitation: FBT emphasizes creating an ecology that supports long-term change, which includes modifying the family environment, reshaping peer networks, & ensuring that there are community resources available to maintain change.
  Interventions: Behavioral: Family-based Behavioral Weight Loss Treatment
- Caregivers: Family-based Behavioral Weight Loss Treatment (FBT) (Experimental): * Traffic Light Eating Plan: All foods are assigned a color of the traffic light depending on their energy density & nutritional quality. Participants are encouraged to set dietary goals to decrease the number of RED food servings consumed daily & to increase the consumption of GREEN & YELLOW foods.
  * Traffic Light Activity Plan: Activities are assigned colors of the traffic light depending on intensity levels. Families are encouraged to increase time spent in GREEN activities and decrease RED activities.
  * Behavior Change Strategies: Behavior modification will be fostered using several different strategies
  * Social Facilitation: FBT emphasizes creating an ecology that supports long-term change, which includes modifying the family environment, reshaping peer networks, & ensuring that there are community resources available to maintain change.
  Interventions: Behavioral: Family-based Behavioral Weight Loss Treatment

INTERVENTIONS:
Behavioral: Family-based Behavioral Weight Loss Treatment — The treatment includes: 1) the Traffic Light Eating Plan; 2) the Traffic Light Activity Program, 3) a variety of behavioral change strategies e.g., stimulus control, self-monitoring, planning, goal setting and 4) facilitation of support in the family and peer environments to optimize the durability and generalizability of health habits across multiple social and environmental contexts
  Other Names: FBT

SUMMARY:
A single-arm, non-randomized four-month trial of the adapted family-based behavioral weight loss treatment (FBT) intervention will be conducted to evaluate its acceptability, feasibility, and preliminary indications of efficacy including measures of relative weight change and associated secondary outcomes (e.g., weight related health behaviors, health related quality of life), among 40 childhood acute lymphoblastic leukemia (ALL) survivors and their families.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking caregiver-child dyads
* Children must be between ages of 5-18
* Child must be overweight or obese (defined as a BMI greater than the 85th percentile for their age and sex)
* Child must have been diagnosed with ALL
* Child must have completed their final cancer treatment and currently be in remission
* Only children and adolescents who have not yet graduated from high school and are living at home with their caregiver at least 50% of the time will be invited to enroll
* Participating caregivers and children must be able to perform some level of exercise

Exclusion Criteria:

* Children who are wards of the state
* Caregivers and/or children who are taking a weight altering medication without being at current dosage for at least six months and weight stable for at least three months
* Caregivers and/or children who are actively involved in another intensive weight loss program
* Caregivers and/or children who have undergone weight loss surgery within the last two years and/or who are still losing weight
* Caregivers and/or children with certain diagnosed psychiatric conditions (e.g., history of/active eating disorder, developmental delays/intellectual disabilities such as Down's syndrome and severe presentations of autism spectrum disorder, active suicidal ideation, psychotic symptoms, manic or hypomanic episodes, severe substance use disorder) that would interfere with their ability to participate
* Caregivers and/or children with certain chronic medical conditions (e.g., type 1 diabetes, muscular dystrophy) for whom participation may be contraindicated

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Acceptability of Family-Based Behavioral Treatment as measured by The Acceptability of Intervention Measure (AIM) | At completion of intervention (estimated to be at 4 months)
  -4 questions about acceptability of the intervention measure. Answers range from completely disagree to completely agree. The higher the score indicates higher acceptability of the intervention measure.
Appropriateness of Family-Based Behavioral Treatment as measured by Intervention Appropriateness Measure (IAM) | At completion of intervention (estimated to be at 4 months)
  -4 questions about appropriateness of the intervention measure. Answers range from completely disagree to completely agree. The higher the score indicates higher appropriateness of the intervention measure.
Acceptability of Family-Based Behavioral Treatment as measured by the Client Satisfaction Questionnaire (CSQ-8) | At completion of intervention (estimated to be at 4 months)
  -8 questions asking about satisfaction of intervention. The CSQ-8 offers four response options for each item (1-4) and an overall score is calculated by summing the respondent's rating score for each item. Scores range from 8-32 with higher scores indicating higher satisfaction.
Feasibility of Family-Based Behavioral Treatment as measured by Feasibility of Intervention Measure (FIM) | At completion of intervention (estimated to be at 4 months)
  -4 questions about feasibility of the intervention measure. Answers range from completely disagree to completely agree. The higher the score indicates higher feasibility of the intervention measure.

SECONDARY OUTCOMES:
Change in relative height (children only) | Baseline, end of intervention (at 4 months), 6 months, and 12 months
Change in dietary intake | Baseline, end of intervention (at 4 months), 6 months, and 12 months
  -Two assisted 24-hour dietary recalls encompassing one weekday and one weekend day and guided by the Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24) will be completed for each participant. This data will be used to measure dietary quality according to the Healthy Eating Index (HEI). The HEI includes a total score as well as sub scores for items such as total fruit intake, whole fruit intake, and total vegetable intake. Total score and sub-scores will be presented.
Change in relative weight | Baseline, end of intervention (at 4 months), 6 months, and 12 months
Change in physical activity as measured by HBSC adaptation | Baseline, end of intervention (at 4 months), 6 months, and 12 months
  -Self- (for children 10+ years) and parent-reported physical activity behavior will be collected via an adapted version of the Health Behavior in School Age Children survey. This three-question survey assesses the amount of time spent on moderate to vigorous physical activity and sedentary behaviors.
Change in physical activity as measured by International Physical Activity Questionnaire (IPAQ) (short) | Baseline, end of intervention (at 4 months), 6 months, and 12 months
  -The IPAQ measures duration and frequency of activity over the past seven days. An overall score can be calculated, as well as sub-scores for moderate- and vigorous-intensity activity

CONTACTS AND LOCATIONS:
Overall Officials: Jessica J Jakubiak, MA, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jakubiak J, Guan M, Khan S, Fowler LA, Bates CR, King AA, Hayashi RJ, Fitzsimmons-Craft E, Wilfley DE. Adaptation of Family-Based Healthy Weight Program for Children who Survived Leukemia. Clin Pract Pediatr Psychol. 2024 Mar;12(1):93-103. doi: 10.1037/cpp0000495. Epub 2023 Oct 5. PMID 38559896
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu